CLINICAL TRIAL: NCT04536259
Title: Assessing People's Hospital Outpatient Appointment Preferences in the United Kingdom
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Warwick (Other)
Responsible Party: Principal Investigator, Kelly Ann Schmidtke, Assistant Professor, University of Warwick
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: BSREC 110/19-20
Record Dates: First submitted 2020-08-24; First posted 2020-09-02 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Hospital Outpatient Clinics; Chronic Disease
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Intervention Model Description: Consenting participants be randomly assigned to one of three groups in a 1:1:1 fashion. Each group will be asked to imagine receiving an invitation to attend a hospital outpatient appointment by video or in-person. In the first group, the proposed attendance mode will be by video. In the second group, the proposed attendance mode will be in-person. In the third group, participants will simply be asked to select which mode of attendance they prefer: video or in-person.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Video Default (Experimental): The case and response options participants in this group will be asked to consider is provided below.
  Imagine that a hospital clinician you have been seeing for over a year tells you that that upon reviewing your patient notes they would like you to attend your next consultation by video.
  Consider each of the response options below, and select the one that best describes how you would respond to your clinician.
  A) Yes, I would be happy to attend a video consultation. B) If possible, I would rather attend the appointment in person.
  Interventions: Behavioral: Video Default
- In-Person Default (Experimental): The case and response options participants in this group will be asked to consider is provided below.
  Imagine that a hospital clinician you have been seeing for over a year tells you that that upon reviewing your patient notes they would like you to attend your next consultation in person.
  Consider each of the response options below, and select the one that best describes how you would respond to your clinician.
  A) Yes, I would be happy to attend an in-person consultation. B) If possible, I would rather attend the appointment by video.
  Interventions: Behavioral: In-Person Default
- Active Choice (Experimental): The case and response options participants in this group will be asked to consider is provided below.
  Imagine that a hospital clinician you have been seeing for over a year tells you that that upon reviewing your patient notes they would like you to attend a consultation by video or in person.
  Consider each of the response options below, and select the one that best describes how you would respond to your clinician.
  A) I would prefer a video consultation. B) I would prefer an in-person consultation.
  Interventions: Behavioral: Active Choice

INTERVENTIONS:
Behavioral: Video Default — The case and response options participants in this group will be asked to consider is provided below.
  Imagine that a hospital clinician you have been seeing for over a year tells you that that upon reviewing your patient notes they would like you to attend your next consultation by video.
  Consider each of the response options below, and select the one that best describes how you would respond to your clinician.
  A) Yes, I would be happy to attend a video consultation. B) If possible, I would rather attend the appointment in person.
  Arms: Video Default
Behavioral: In-Person Default — The case and response options participants in this group will be asked to consider is provided below.
  Imagine that a hospital clinician you have been seeing for over a year tells you that that upon reviewing your patient notes they would like you to attend your next consultation in person.
  Consider each of the response options below, and select the one that best describes how you would respond to your clinician.
  A) Yes, I would be happy to attend an in-person consultation. B) If possible, I would rather attend the appointment by video.
  Arms: In-Person Default
Behavioral: Active Choice — The case and response options participants in this group will be asked to consider is provided below.
  Imagine that a hospital clinician you have been seeing for over a year tells you that that upon reviewing your patient notes they would like you to attend a consultation by video or in person.
  Consider each of the response options below, and select the one that best describes how you would respond to your clinician.
  A) I would prefer a video consultation. B) I would prefer an in-person consultation.
  Arms: Active Choice

SUMMARY:
The sustainability of the United Kingdom's National Health Service's (NHS) is threatened immediately by Covid-19 and continually by an increasing prevalence of long-conditions that cannot be cured but can be maintained. Shifting traditional face-to-face outpatient appointments to remote video consultations may help the NHS continue to serve patients efficiently. While much research has examined healthcare providers' attitudes and beliefs about remote video consultations, less has attempted to understand how NHS service providers should invite patients to attend them. The present study examines how the framing of an invitation to attend a hospital outpatient appointment by video influences the proportion of people who agree to attend by video. It also explores some of the barriers and facilitators people may experience to attending appointments by video across diagnostic complexities and age groups. The results of this study should help hospitals better present patients with the option to attend video consultations where appropriate, and provide support to mitigate common barriers to people's willingness to give video consultations a go.

ELIGIBILITY:
Inclusion Criteria:

All participants will:

* be 18 years old or older;
* be resident in the United Kingdom; and
* indicate having been diagnosed with a chronic diseases such as diabetes, heart disease, stroke etc.

Exclusion Criteria:

* be less than 18 years old;
* not be resident in the United Kingdom; and
* not indicate having been diagnosed with a chronic diseases such as diabetes, heart disease, stroke etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1481 (Actual)
Dates: Start 2020-09-11 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Response to the outpatient invitation | One day
  Participants responses will indicate whether they would prefer a video or in-person appointment.

CONTACTS AND LOCATIONS:
Overall Officials: Kelly A Schmidtke, PhD, Principal Investigator — University of Warwick
Locations (1):
- Kelly Schmidtke, Coventry, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The anonymised individual level data may be made available upon reasonable request within 10 years of the project being published in an academic jourhnal or may be published with an article if required by the journal.